CLINICAL TRIAL: NCT00003412
Title: Phase I Study of Post Transplant rhIL-12 High Dose Cyclophosphamide, Thiotepa, and Carboplatin in the Treatment of Metastatic Breast Carcinoma
Brief Title: Interleukin-12 in Treating Women With Metastatic Breast Cancer Who Have Received High-Dose Chemotherapy and Peripheral Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066424; BIH-L97-0252; NCI-T98-0002
Record Dates: First submitted 1999-11-01; First posted 2004-03-31 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2001-10

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Interleukin-12 Subunit p35

INTERVENTIONS:
Biological: recombinant interleukin-12

SUMMARY:
RATIONALE: Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill breast cancer cells.

PURPOSE: Phase I trial to study the effectiveness of interleukin-12 in treating women with metastatic breast cancer who have received high-dose chemotherapy and peripheral stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxic effect profile and maximum tolerated dose of interleukin-12 (rhIL-12) in women with advanced breast cancer who have undergone high dose chemotherapy with stem cell rescue. II. Determine the effect of rhIL-12 on cellular and humoral immune systems following high dose chemotherapy. III. Explore the effect on treatment failure of rhIL-12 after high dose chemotherapy with stem cell rescue.

OUTLINE: This is a dose escalation study of interleukin-12 (rhIL-12). RhIL-12 therapy begins 3-5 weeks after discharge from the chemotherapy/stem cell transplant hospitalization or 2-3 weeks after completion of posttransplant radiation. Patients receive rhIL-12 subcutaneously twice a week for 12 consecutive weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients are treated at each dose level of rhIL-12. The maximum tolerated dose is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicity. Patients are followed every 2 months after treatment.

PROJECTED ACCRUAL: Approximately 6-35 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IV breast cancer presenting as primary metastatic disease or with recurrence after an initial diagnosis of localized disease Enrollment in protocol for high dose chemotherapy with stem cell rescue using the "STAMP V" regimen (cyclophosphamide, thiotepa, and carboplatin) No enrollment in research transplant protocol whose primary endpoint is response duration or recovery time from toxic effects No brain or CNS metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 to 60 Sex: Female Menopausal status: Not specified Performance status: Karnofsky 80-100% Life expectancy: At least 6 months Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT no greater than 2.5 times normal Renal: Creatinine no greater than 1.8 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: Systolic ejection fraction at least 50% No significant cardiovascular disease or cardiac arrhythmia requiring drug or device intervention Pulmonary: DLCO and FEV1 greater than 50% Neurologic: No significant peripheral neuropathy or CNS disease Other: Fertile patients must use effective contraception Not pregnant or lactating Not HIV positive No concurrent active infections requiring IV antibiotic therapy No significant gastrointestinal bleeding or uncontrolled peptic ulcer disease No history of inflammatory bowel disease No clinically significant autoimmune disease No other serious illness or medical condition

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics No concurrent chemotherapy Endocrine therapy: No concurrent corticosteroids Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: At least 4 weeks since any investigational drugs No concurrent investigational drugs

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States